CLINICAL TRIAL: NCT00624247
Title: Early Versus Delayed Routine HIV Testing in Connecticut Jails
Acronym: SWAB
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 0705002664
Record Dates: First submitted 2008-02-18; First posted 2008-02-27 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: routine HIV testing; jails; criminal justice system; substance abuse; mental illness; HIV
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Immediate (Other): Individuals assigned to be approached for routine HIV testing immediately upon admission to the jail.
  Interventions: Other: routine HIV testing
- Following Day (Other): Individuals assigned to be approached for routine HIV testing the day following admission to the jail.
  Interventions: Other: routine HIV testing
- Delayed (Other): Individuals assigned to be approached for routine HIV testing several days following admission to the jail.
  Interventions: Other: routine HIV testing

INTERVENTIONS:
Other: routine HIV testing — Potential subjects are offered swabbing as part of HIV testing by jail medical staff or study staff. All potential subjects are told HIV results can now be made available within a short period of time using an oral swab. Anyone not wanting HIV test results is allowed to refuse at the time of offering the HIV test and not be swabbed. If the inmate agrees to be swabbed and tested, he or she then meets with a member of the research study staff who discusses two separate informed consents - one for study participation and one for HIV testing.

SUMMARY:
The objective of this non-randomized, controlled, trial is to evaluate the optimal time to approach newly incarcerated jail inmates for routine opt-out HIV testing in a manner that maximizes the number of individuals able to demonstrate capacity to consent and willingness to receive HIV testing.

DETAILED DESCRIPTION:
Primary outcome: proportion of individuals in each assigned group that agree to be swabbed for HIV testing and are able to consent to the study.

The prevalence of HIV infection in the United States is four times greater in correctional settings compared to the general population. Because prisons and jails house a population facing a disproportionate share of the burden of HIV infection, these facilities serve as important sites for the testing and treatment of HIV. The Center for Disease Control and Prevention's recent recommendations to implement routine opt-out HIV testing in all healthcare settings presents an important challenge and opportunity to correctional institutions. By effectively implementing routine opt-out testing, correctional facilities can expand HIV testing to one of society's most at-risk populations. Subsequently, testing can lead to appropriate access to counseling and treatment both within the correctional setting and upon release into the community.

Although jails interact with a larger number of individuals at risk for HIV infection than do prisons, they also pose unique logistical and health-related constraints in several important ways that impact HIV testing strategies. Jail populations experience short periods of incarceration and high rates of turnover with many-fold greater admissions and discharges. Jails also house individuals with higher rates of acute intoxication from psychoactive drugs, uncontrolled mental illness, and suicidal behavior. The suicide rate in jails is three times that in state prisons; nearly a quarter of these suicides take place within the first 48 hours of admission. Furthermore, the individuals who enter jails have higher recent risk behaviors for HIV than those in prisons.

Given these considerations, a major challenge to implementing routine opt-out HIV testing in jails is choosing the optimal time to conduct testing. The timing of delivering non-emergent, traumatically emotional health information (such as a preliminary positive result in an asymptomatic patient) must be carefully considered. Recently incarcerated inmates might be too intoxicated or psychologically distressed to demonstrate capacity to consent to or opt out of routine testing, and may be unprepared to consider and respond to the consequences of a preliminary positive HIV test result. Likewise, the challenge with postponing testing is that many individuals experience very short stays in jail, with approximately one-third leaving within 48 hours, followed by further attrition daily for the first week and may lose the opportunity for getting life-saving information in a timely manner.

Therefore, the objective of this study is to evaluate the optimal time to approach newly incarcerated jail inmates for routine opt-out HIV testing in a manner that maximizes the number of individuals able to demonstrate capacity to consent and willingness to receive HIV testing.

ELIGIBILITY:
Inclusion Criteria:

* All newly incarcerated inmates will be eligible for this study.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The proportion of individuals in each testing group who are orally swabbed and consented to rapid HIV testing. | Immediately, the following evening, and 7 days post-entry

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, MD, Principal Investigator — Yale University AIDS Program
Locations (2):
- United States (2):
  - New Haven Community Correctional Center, New Haven, Connecticut
  - York Correctional Institution, Niantic, Connecticut

REFERENCES:
- [Background] Kavasery R, Maru DS, Sylla LN, Smith D, Altice FL. A prospective controlled trial of routine opt-out HIV testing in a men's jail. PLoS One. 2009 Nov 25;4(11):e8056. doi: 10.1371/journal.pone.0008056. PMID 19946371
- [Background] Kavasery R, Maru DS, Cornman-Homonoff J, Sylla LN, Smith D, Altice FL. Routine opt-out HIV testing strategies in a female jail setting: a prospective controlled trial. PLoS One. 2009 Nov 25;4(11):e7648. doi: 10.1371/journal.pone.0007648. PMID 19946370